CLINICAL TRIAL: NCT02577081
Title: Assessment of the Risk of Contralateral Non Simultaneous Neck of Femur Fracture in the Elderly. CT Based Study.
Brief Title: Assessment of the Risk of Contralateral Non Simultaneous Neck of Femur Fracture in the Elderly.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, niv marom, Niv marom, Resident, Department of Orthopaedic surgery, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0163-15-MMC
Record Dates: First submitted 2015-09-24; First posted 2015-10-16 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Neck of Femur Fracture
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAT scan (Experimental): A CAT scan will be done for all participants. The scan will include the pelvis and 2 femurs.
  Interventions: Other: CAT scan (CT scan)

INTERVENTIONS:
Other: CAT scan (CT scan) — all patients will pass a CAT scan of ths pelvis and the 2 femurs. No other interventions are required.

SUMMARY:
Neck of femur fractures are common in the elderly and are the source of significant morbidity and mortality. This study is based on a new technique developed in Ben Gurion University, with which investigators are able to asses the structural 3 dimensional strength of a bone by applying a unique simulation on a CAT scan of the bone. The purpose of this study is to evaluate the risk of a contralateral neck of femur fracture after the first neck of femur fracture and to estimate the potential fracture characteristics.

DETAILED DESCRIPTION:
Neck of femur fractures are common in the elderly and are the source of significant morbidity and mortality. literature shows that around 10 percent of those who fracture their femoral neck for the first time will later fracture their contralateral neck of femur and in most cases with the same fracture characteristics. This study is based on a new technique developed in Ben Gurion University, with which investigators are able to asses the structural 3 dimensional strength of a bone by applying a unique simulation on a CAT scan of the bone. The purpose of this study is to evaluate the risk of a contralateral neck of femur fracture after the first neck of femur fracture and to estimate the potential fracture characteristics.

ELIGIBILITY:
Inclusion Criteria:

* 70-90 years old patients admitted to the orthopaedic department after neck of femur fracture.
* No contra lateral femur pathology.
* Consent for pelvis and femurs CAT scan.

Exclusion Criteria:

* Known pathology in other lower limbs joints in the body.
* History of previous fractures or operations in lower limbs.

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The risk of a contralateral neck of femur fracture | 5 years
  A patient specific analysis based on CT scan and finite element analysis will be done on both neck of femurs.

SECONDARY OUTCOMES:
3 dimensional charataristics of the neck of femur fracture | 1 year
  The CAT scan will provide 3 dimensional characteristics of the current neck of femur fracture as well as the predicted one in the contralateral femur. The fracture will be described using orthopaedic classifications, such as: garden classification for neck of femur fractures and AO classification for intertrochanteric fractures of the femur.

CONTACTS AND LOCATIONS:
Overall Officials: niv marom, MD, Study Chair — meir medical cenrter
Locations (1):
- Meir medical center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaumetou E, Zilber S, Hernigou P. Non-simultaneous bilateral hip fracture: epidemiologic study of 241 hip fractures. Orthop Traumatol Surg Res. 2011 Feb;97(1):22-7. doi: 10.1016/j.otsr.2010.07.011. Epub 2011 Jan 15. PMID 21239241
- [Background] Burgers PT, Zielinski SM, Mailuhu AK, Heetveld MJ, Verhofstad MH, Roukema GR, Patka P, Poolman RW, Van Lieshout EM; Dutch femoral neck fracture investigator group. Cumulative incidence and treatment of non-simultaneous bilateral femoral neck fractures in a cohort of one thousand two hundred and fifty patients. Int Orthop. 2014 Nov;38(11):2335-42. doi: 10.1007/s00264-014-2447-2. Epub 2014 Aug 3. PMID 25086819
- [Background] Yosibash Z, Trabelsi N, Milgrom C. Reliable simulations of the human proximal femur by high-order finite element analysis validated by experimental observations. J Biomech. 2007;40(16):3688-99. doi: 10.1016/j.jbiomech.2007.06.017. Epub 2007 Aug 13. PMID 17706228
- [Background] Yosibash Z, Tal D, Trabelsi N. Predicting the yield of the proximal femur using high-order finite-element analysis with inhomogeneous orthotropic material properties. Philos Trans A Math Phys Eng Sci. 2010 Jun 13;368(1920):2707-23. doi: 10.1098/rsta.2010.0074. PMID 20439270
- [Background] Trabelsi N, Yosibash Z, Wutte C, Augat P, Eberle S. Patient-specific finite element analysis of the human femur--a double-blinded biomechanical validation. J Biomech. 2011 Jun 3;44(9):1666-72. doi: 10.1016/j.jbiomech.2011.03.024. Epub 2011 Apr 15. PMID 21497354